CLINICAL TRIAL: NCT03384927
Title: Effect of Treatment Dairy on Botulinum Toxin Treatment for Muscle Overactivity (Spasticity). A Randomised Cross-over Study.
Brief Title: Effect of Treatment Dairy for Spasticity
Status: Enrolling by invitation | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Bo Biering-Soerensen, Doctor, Head of Clinic for spasticity, Rigshospitalet, Denmark
Other Study IDs: RH-2017-292
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Spasticity, Muscle
Keywords: Treatment diary
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
1. Assessing whether the treatment diary can help optimize the overall treatment of patients.
2. To assess whether the patient finds the treatment diary useful and worth spending time on. Also if the patient finds it easier to evaluate the treatment and, if necessary, set new goals.
3. To assess whether the patient's quality of life is increased by the use of the treatment diary.

DETAILED DESCRIPTION:
Hypothesis:

A treatment diary will increase the patient's awareness of which spasticity symptoms are significant and can enable the patients to evaluate the treatment more easily.

This will result in more relevant treatment goals. At the same time the treatment can be better addressed to the individual patient at routine controls. In addition, the treatment diary will result in closer cooperation between the physiotherapists and occupational therapists and the physician who administers the botulinum toxin. This collaboration is expected to lead to better common goals and optimization of treatment.

Finally, it is expected that the above will help to increase the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received at least two previous treatments before inclusion, ie. with approx. 3 months apart, and it is assessed that the patients have good effect of the treatments in relation to the agreed treatment goals.

Exclusion Criteria:

* Patients where changes are planned regarding their treatment for muscle overactivity during the study period.

Patients where the disease is not stable and where it may have a major influence on the treatment effect of botulinum toxin treatment during the study period and where it can be difficult to set SMART (Specific, Measurable, Accepted, Realistic, Timed) goals.

Patients who have previously been treated and have used a treatment diary in connection with the botulinum toxin treatment.

Patients who can not collaborate on completing goals and evaluating treatment effect due to language or cognitive problems.

Patients who at the same time are being treated with botulinum toxin in the bladder.

If significant changes occur in the patient's health, which may involve new cancer, stroke, multiple sclerosis attack, etc. during the study period, the participant will be withdrawn from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with muscle overactivity / spasticity independent of the cause and who are being followed as outpatients in the Spasticity Clinic, Neurological Clinic, Rigshospitalet Glostrup.
Sampling Method: Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2017-12-11 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient becomes more satisfied with their treatment using the treatment diary | October 2019
  To assess if the patient becomes more satisfied with their treatment using the treatment diary. This is assessed by a change in the score on the treatment assessment questionnaire (Questionnaire 1).

SECONDARY OUTCOMES:
To assess if the patient's quality of life is improved using the treatment diary. | October 2019
  To assess if the patient's quality of life is improved using the treatment diary. This is assessed by a change in the score on the quality of life, SF-12 (Questionnaire 2)
The patients' assessment of the treatment diary will be described (Questionnaire 3). | October 2019
  the patients' assessment of the treatment diary will be described (Questionnaire 3).

CONTACTS AND LOCATIONS:
Overall Officials: Bo BS Biering-Soerensen, Doctor, Principal Investigator — Spasticity Clinic, Rigshospitalet Glostrup
Locations (1):
- Spasticity Clinic, Neurological Clinic, Rigshospitalet Glostrup, Glostrup Municipality, Denmark